CLINICAL TRIAL: NCT07188376
Title: Mitigating the Disinhibiting Effects of Alcohol With Transcranial Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael J. Wesley, PhD (Other)
Responsible Party: Sponsor-Investigator, Michael J. Wesley, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 106047
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Risk Behaviors
Keywords: TMS; Impulsivity
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: Each participant completes all five conditions (Alcohol + iTBS, Alcohol + cTBS, Placebo + iTBS, Placebo + cTBS, and Alcohol + sham)
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a study with five experimental conditions that are combinations of alcohol (real, placebo) and brain stimulation (real and sham). The participant will be blinded to all alcohol conditions (alcohol = single blind). The participant and experimenter will be blinded to the brain stimulation condition (TMS = double blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active alcohol (Experimental): Participants consume a real alcoholic beverage (ethanol diluted 1:3 with soda, consumed over 10 minutes) designed to produce a peak BAC of ~0.08%
  Each session includes baseline task performance, TMS delivered at estimated peak blood alcohol concentration, and follow-up testing to assess changes in impulsivity. This within-subject crossover design allows each participant to serve as their own control to isolate TMS effects.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Transcranial Magnetic Stimulation
- Placebo alcohol (Placebo Comparator): Participants consume a placebo beverage matched in volume and appearance to the alcoholic beverage, but without an intoxicating dose (soda with alcohol misted on top to simulate scent, consumed over 10 minutes).
  Each session includes baseline task performance, TMS delivered at estimated peak blood alcohol concentration, and follow-up testing to assess changes in impulsivity. This within-subject crossover design allows each participant to serve as their own control to isolate TMS effects.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — Intermittent Theta Burst Stimulation (iTBS) is then delivered to the left DLPFC using a MagVenture TMS device. Each iTBS session includes 600 pulses delivered in 3-pulse bursts at 50 Hz, every 200 ms (5 Hz), in 2 sec on / 8 sec off cycles at 110% resting motor threshold (RMT). Stimulation is ramp-up from 80% to 110% RMT (~90 pulses). Two iTBS sessions are given per visit, separated by 30 minutes. The second session is timed to correspond to the peak BAC.
Device: Continuous Theta Burst Stimulation — Continuous Theta Burst Stimulation (cTBS) is then delivered to the left DLPFC using a MagVenture TMS device. Each cTBS session includes 2 bouts of 1800 pulses separated by a 1 minute rest period. Each bout is delivered in 3-pulse bursts at 50 Hz, every 200 ms (5 Hz), continuously for ~120 seconds at 110% resting motor threshold (RMT). Stimulation is ramped up from 80% to 110% RMT over the first 30 seconds. Two cTBS sessions are given per visit, separated by 30 minutes. The second session is timed to correspond to the peak BAC.
Device: Sham Transcranial Magnetic Stimulation — Sham Transcranial Magnetic Stimulation (TMS) is delivered to the left DLPFC using the sham side of a MagVenture TMS coil, paired with synchronized scalp electrodes to mimic the sensation of real TMS. The sham procedure matches the timing and auditory cues of either iTBS or cTBS protocols, depending on random assignment. Two sham stimulation sessions are given per visit, separated by 30 minutes. The second session is timed to correspond to the peak BAC.
  Arms: Active alcohol

SUMMARY:
The goal of this clinical trial is to learn how a specific type of brain stimulation affects alcohol-related decision-making and self-control in adults who drink alcohol. The main questions the study aims to answer are:

* Does brain stimulation change how people behave after drinking alcohol?
* Does the combination of alcohol and different types of brain stimulation affect people's ability to make thoughtful decisions or resist impulses?

Researchers will compare the effects of two types of brain stimulation, intermittent theta burst stimulation (iTBS) and continuous theta burst stimulation (cTBS), after people drink alcohol or a placebo drink. A sham (placebo) stimulation condition will also be included. The study uses a within-person design, which means each participant will take part in all conditions.

Participants will:

* Attend five separate study visits
* Drink either an alcoholic or placebo beverage
* Receive one of the brain stimulation conditions (real or sham)
* Complete decision-making tasks before and after drinking

The tasks will measure things like impulsive choices and reaction time. The researchers hope this study will help identify how brain stimulation could be used to improve decision-making during intoxication, which might one day reduce harmful drinking behaviors or prevent alcohol-related accidents.

DETAILED DESCRIPTION:
This study aims to understand how brain stimulation affects decision-making and behavioral control after alcohol consumption. Many harmful events related to alcohol use are the result of impaired decision-making while intoxicated. Although there are medications that reduce alcohol cravings, there are few tools available to reduce the negative behavioral effects of alcohol once someone has already consumed it.

This clinical trial uses non-invasive brain stimulation, known as transcranial magnetic stimulation (TMS), to target a brain area called the prefrontal cortex, which helps regulate decision-making and self-control. TMS can increase or decrease activity in targeted brain areas using magnetic pulses. Two specific types of stimulation will be tested:

* iTBS (intermittent theta burst stimulation): typically increases brain activity
* cTBS (continuous theta burst stimulation): typically decreases brain activity

Participants will be healthy adults who report regularly drinking alcohol. Each participant will attend five sessions in a randomized, within-subject design. Across the sessions, participants will experience each of the following conditions:

1. Alcohol + iTBS
2. Alcohol + cTBS
3. Placebo drink + iTBS
4. Placebo drink + cTBS
5. Alcohol + sham (placebo) stimulation

Each session will be conducted on a separate day and will include:

* A baseline set of tasks (before drinking or stimulation)
* Drinking either an alcoholic or placebo beverage
* TMS delivered during the rise and peak of blood alcohol concentration
* A second round of behavioral tasks administered at peak intoxication and again during the descending limb of the blood alcohol curve

The behavioral Go/No-Go Task will measure:

- How well participants can stop themselves from making automatic responses

The study's goals are to:

* Test whether brain stimulation can reduce impulsive behaviors under the influence of alcohol
* Understand the separate and combined effects of alcohol and TMS on decision-making
* Identify which type of TMS is most effective in modulating intoxicated behavior

The stimulation dose and session timing are designed to align with the typical rise and fall of blood alcohol levels. Each stimulation session will use a "ramping" protocol to gradually increase stimulation intensity, improving tolerability. Safety and tolerability will be carefully monitored.

This study builds on previous work showing that TMS can influence decision-making but is the first to examine whether TMS can be used during alcohol intoxication to improve behavioral control. If successful, the findings may lead to new interventions for preventing risky or harmful behaviors associated with alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-29
* Must be competent in English
* BMI between 19 and 26
* At least a high school education
* Moderate alcohol users (e.g., at least occasional alcohol use, without meeting criteria for alcohol use disorder)
* Negative urine drug screen for illicit drugs
* Negative urine pregnancy test (if applicable) on testing days

Exclusion Criteria:

* History of seizures or a first-degree relative with seizure history
* History of head trauma or other CNS injuries
* Current or past psychiatric disorders (including substance use disorder, except nicotine or caffeine)
* Contraindications for non-invasive brain stimulation (e.g., metal implants, pacemaker)
* Currently pregnant or breastfeeding
* Current use of medications that lower seizure threshold
* Positive alcohol withdrawal symptoms
* Smokes more than five cigarettes per day (to avoid acute nicotine effects or withdrawal during visits)

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Inhibition Failures (p-failures) | Measured at baseline, immediately after the second TMS session at peak BAC (~0.08%), and again on the descending limb of BAC (~0.05%) (approximately 3 hours total)
  Change in the proportion of inhibition failures (p-failures) on the cued Go/NoGo task from baseline to post-intervention under each experimental condition. Higher p-failure rates reflect poorer inhibitory control. This outcome will be measured following each TMS and alcohol condition (iTBS, cTBS, sham × active or placebo alcohol), and assessed across timepoints (peak Blood Alcohol Concentration (BAC) ~0.08% and descending BAC ~0.05%).

SECONDARY OUTCOMES:
Reaction Time on Go Trials | Measured at baseline, at peak BAC, and on the descending limb of BAC (approximately 3 hours total)
  Average response latency (in milliseconds) to correctly identified Go stimuli on the cued Go/NoGo task. This measure reflects psychomotor speed and processing efficiency and will be used to assess general effects of alcohol and/or TMS interventions.
Change in Blood Alcohol Concentration-related Task Performance | Assessed within-session at peak and descending BAC (approximately 3 hours total)
  Exploratory analysis of behavioral changes (e.g., p-failures, Go reaction times) across different phases of the blood alcohol curve (peak ~0.08% vs. descending ~0.05%) under each intervention condition. This outcome will assess whether effects of TMS on inhibitory control and response latency are state-dependent relative to the intoxication curve.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wesley, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided